CLINICAL TRIAL: NCT03998267
Title: Qatar Diabetes Mobile Application Trial
Acronym: QDMAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Collaborators: Qatar Computing Research Institute (QCRI) (Unknown); Droobi Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17292
Record Dates: First submitted 2019-06-11; First posted 2019-06-26 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Type2 Diabetes Mellitus
Keywords: mobile health; m-health
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Subjects with T2DM will be randomised into an intervention arm and standard care arm. Subjects in the intervention arm receive usual diabetes care in addition to the mobile app while subjects in the standard care will receive usual diabetes care only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Active Comparator): For the subjects using the app (intervention group): The mobile app team shall do the following:
  * Educate/train patients on app usage
  * Patients will be subscribed to the app and their profile on the app will be created
  * Subjects will log in their blood sugar readings and communicate with the mobile app team (educators and physician) via the app
  * Additionally patients will be placed on a diet and lifestyle plan as agreed upon by the patient and health care provider team, best suited towards the patient's needs
  * Throughout the study, patient will receive notifications and advice on how to follow diet and lifestyle changes
  * Throughout the study; patient interaction and app usage will be tracked
  * Patients will additionally be interviewed by the research team together with Droobi to capture app experience at 3 months and 6 months
  Interventions: Device: Droobi; Other: Standard of care
- Standard of care arm (Placebo Comparator): For the subjects not using the app (the standard of care group):
  * At time 0, will be seen by the dietician and diabetes educators at HGH endocrine clinics as part of standards of care
  * The educators contact number and diabetes hotline number will be provided to the patients
    o The diabetes hotline number #16099 is a new service provided to diabetes patients at the national diabetes center to help communicate with the diabetes educators with questions relating to their diabetes management, medication adjustment such as dose titrations etc.
  * Appointments thereafter with the educator and/or dietician will be decided and scheduled according to the individual patient needs, with a minimum visit every 3 months during the study period
  Interventions: Other: Standard of care

INTERVENTIONS:
Device: Droobi — A new mobile application, specifically built for the diabetes patients in Qatar with the help of local expertise.
  Arms: Intervention arm
Other: Standard of care — Standard of care including physicians, dietetics and diabetes educators support

SUMMARY:
Diabetes mobile technology is an emerging and rapidly expanding field that seeks to combine cutting edge behavioral insights with best practice in diabetes self management education to improve patient empowerment and deliver better patient outcomes.The question that arises is whether or not, diabetes mobile applications are effective in improving glycemic control, clinical outcomes, quality of life and overall patient satisfaction, in diabetic patients in Qatar. To answer this, we plan to enroll 90 diabetic patients into a custom-made diabetes app for Qatar (Droobi) (as intervention group) in comparison with 90 diabetic patients followed in the current standard care, matched in characteristics (as control group). We have the hypothesis that with utilization of the mobile application, patients will have improved glycemic control, improved self management and patient empowerment; together with improved patient-educator/doctor interaction.

ELIGIBILITY:
Inclusion Criteria:

* • Adults with T2DM (more than 18 yrs of age and younger than 60) who are able to provide consent

  * Arabic speaking and non-arabic speaking T2DM patients, who can communicate in Arabic and or English language.
  * Uncontrolled diabetes with HbA1c more than or equal to 8.5%
  * T2DM on insulin with or without any other oral medication
  * Subject must have a smart phone (must be an iOS (Apple) phone user) and must be interested in using a smart phone app.
  * Subject must have no visual impairment.
  * Minimal level of literacy (able to read and write in english or arabic).
  * To be able to communicate via chat with the mobile app team through the app as evidenced by at least weekly use of any of the social media such as WhatsApp, Viber, Facebook Messenger etc
  * Subject must be willing to utilize a mobile application for diabetes control

Exclusion Criteria:

* • Recent history (3 months) of stroke or Myocardial infarction.

  * Patients with proliferating retinopathy
  * Patients with an acute illness during the past 2 weeks.
  * Patients who plan to be away for more than 3 months.
  * Patients with CKD requiring dialysis.
  * Hypoglycemia unawareness.
  * More than one episode of severe hypoglycemia in the previous 6 months.
  * Female patients who are planning for pregnancy in the coming 6 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-08-22 (Actual); Primary Completion 2020-08-17 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in mean HbA1c | 6 months
  Difference in mean HbA1C between the intervention arm and the standard care
Difference in mean HbA1c | 3 months
  Difference in mean HbA1C between the intervention arm and the standard care

SECONDARY OUTCOMES:
Subject perceptions of diabetes self management | 6 months
  Within subject changes in perceptions of diabetes self-management as assessed by diabetes self-management questionnaire (DSMQ) scores subsection glucose management and overall rating. DSM-Q is a 16 item questionnaire to assess self-care activities associated with glycemic control. Four subscales, 'Glucose Management' (GM), 'Dietary Control' (DC), 'Physical Activity' (PA), and 'Health-Care Use' (HU), as well as a 'Sum Scale' (SS) as a global measure of self-care. Scale scores are calculated as sums of item scores and then transformed to a scale ranging from 0 to 10 (raw score / theoretical maximum score * 10. A transformed score of ten thus represents the highest self-rating of the assessed behavior
Change in subjects attitudes towards disease | 6 months
  Within subject changes in attitudes towards disease assessed the proportion of subjects with diabetes distress scales (DDS) scores consistent with moderate or high distress.The DDS yields a total distress score plus 4 subscale (emotional burden,physical distress, regimen distress and interpersonal distress) scores each addressing a different kind of distress. A mean item score 2.0-2.9 is considered moderate distress and a mean score of more than or equal to 3 is considered high stress.
Changes in insulin doses | 6 months
  Difference in number of recommended insulin dose adjustments per subject between intervention and usual care arm
Changes in reported hypoglycemia | 6 months
  Difference in the number of reported hypoglycemic events per subject between the intervention and usual care arm.
Time to achieve normoglycemia | 6 months
  Reduction in the time required to reach normoglycemia (in-range blood glucose readings) between the intervention and control groups.
Number of clinical interactions | 6 months
  • Differences in the number of clinical interactions per subjects with healthcare providers through the mobile app and through usual means in the standard care
Missed clinical appointments | 6 months
  Percent of missed clinical appointments in each arm.
Weight | 6 months
  Changes in weight from baseline at 6 months
Blood Pressure | 6 months
  Changes in blood pressure from baseline at 6 months
Lipids | 6 months
  Changes in lipids from baseline at 6 months

OTHER OUTCOMES:
Exploratory outcome | 6 months
  Increased mobile application usability by the system usability scale (SUS) at 6 months. It consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree. The participant's scores for each question are converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. An SUS score above a 68 would be considered above average and anything below 68 is below average, however the best way to interpret the results involves "normalizing" the scores to produce a percentile ranking
Exploratory outcome | 6 months
  Increased mobile application acceptance by documentation of patients experiences with the mobile application
Exploratory outcome | 6 months
  Reduction in hospital admissions

CONTACTS AND LOCATIONS:
Overall Officials: Noor N Suleiman, MD, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Hamad General Hospital, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alotaibi MM, Istepanian R, Philip N. A mobile diabetes management and educational system for type-2 diabetics in Saudi Arabia (SAED). Mhealth. 2016 Aug 24;2:33. doi: 10.21037/mhealth.2016.08.01. eCollection 2016. PMID 28293606
- [Background] Cui M, Wu X, Mao J, Wang X, Nie M. T2DM Self-Management via Smartphone Applications: A Systematic Review and Meta-Analysis. PLoS One. 2016 Nov 18;11(11):e0166718. doi: 10.1371/journal.pone.0166718. eCollection 2016. PMID 27861583
- [Background] Seto E, Istepanian RS, Cafazzo JA, Logan A, Sungoor A. UK and Canadian perspectives of the effectiveness of mobile diabetes management systems. Annu Int Conf IEEE Eng Med Biol Soc. 2009;2009:6584-7. doi: 10.1109/IEMBS.2009.5333998. PMID 19964700
- [Background] Kitsiou S, Pare G, Jaana M, Gerber B. Effectiveness of mHealth interventions for patients with diabetes: An overview of systematic reviews. PLoS One. 2017 Mar 1;12(3):e0173160. doi: 10.1371/journal.pone.0173160. eCollection 2017. PMID 28249025
- [Background] Istepanian RS, Zitouni K, Harry D, Moutosammy N, Sungoor A, Tang B, Earle KA. Evaluation of a mobile phone telemonitoring system for glycaemic control in patients with diabetes. J Telemed Telecare. 2009;15(3):125-8. doi: 10.1258/jtt.2009.003006. PMID 19364893
- [Background] Ristau R, Yang J, White J. Evaluation and Evolution of Diabetes Mobile Applications: Key Factors for Health Care Professionals Seeking to Guide Patients.
- [Background] Bonoto BC, de Araujo VE, Godoi IP, de Lemos LL, Godman B, Bennie M, Diniz LM, Junior AA. Efficacy of Mobile Apps to Support the Care of Patients With Diabetes Mellitus: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. JMIR Mhealth Uhealth. 2017 Mar 1;5(3):e4. doi: 10.2196/mhealth.6309. PMID 28249834
- [Background] Alhuwail D. Diabetes Applications for Arabic Speakers: A Critical Review of Available Apps for Android and iOS Operated Smartphones. Stud Health Technol Inform. 2016;225:587-91. PMID 27332269
- [Background] Polonsky WH, Fisher L, Earles J, Dudl RJ, Lees J, Mullan J, Jackson RA. Assessing psychosocial distress in diabetes: development of the diabetes distress scale. Diabetes Care. 2005 Mar;28(3):626-31. doi: 10.2337/diacare.28.3.626. PMID 15735199
- [Background] Schmitt A, Gahr A, Hermanns N, Kulzer B, Huber J, Haak T. The Diabetes Self-Management Questionnaire (DSMQ): development and evaluation of an instrument to assess diabetes self-care activities associated with glycaemic control. Health Qual Life Outcomes. 2013 Aug 13;11:138. doi: 10.1186/1477-7525-11-138. PMID 23937988
- [Derived] Suleiman N, Alkasem M, Al Amer Z, Salameh O, Al-Thani N, Hamad MK, Baagar K, Abdalhakam I, Othman M, Dughmosh R, Al-Mohanadi D, Al Sanousi A, Bashir M, Chagoury O, Taheri S, Abou-Samra AB. Qatar Diabetes Mobile Application Trial (QDMAT): an open-label randomised controlled trial to examine the impact of using a mobile application to improve diabetes care in type 2 diabetes mellitus-a study protocol. Trials. 2022 Jun 16;23(1):504. doi: 10.1186/s13063-022-06334-5. PMID 35710428
- See also: Droobi Health application website — https://www.droobihealth.com/